CLINICAL TRIAL: NCT06904248
Title: Evaluation of the Efficacy and Safety of Meloxicam Injection for Postoperative Analgesia in Abdominal Surgery Patients: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 3 Clinical Trial
Brief Title: Efficacy and Safety of Intravenous Meloxicam in Subjects With Moderate-to-severe Pain Following Abdominal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yangtze River Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YZJ-MLXK-YZ-2208
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Participants With Acute Moderate to Severe Pain Following Abdominal Surgery
MeSH Terms: interventions — Meloxicam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meloxicam Injection (Experimental)
  Interventions: Drug: Meloxicam Injection
- Placebo (Placebo Comparator)
  Interventions: Drug: Sodium Chloride Injection

INTERVENTIONS:
Drug: Meloxicam Injection — Intravenous meloxicam Injection, 30mg every 24 hours, for a total of 2 doses
  Arms: Meloxicam Injection
Drug: Sodium Chloride Injection — Intravenous Sodium Chloride Injection, 18mg every 24 hours, for a total of 2 doses
  Arms: Placebo

SUMMARY:
This study aims to evaluate the analgesic efficacy and safety of meloxicam injection in subjects with moderate-to-severe pain following abdominal surgery. The primary efficacy endpoint is the summed pain intensity difference over 24 hours ( SPID24)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 75 years of age, inclusive.
2. Be scheduled to undergo abdominal surgery under general anesthesia with anticipated moderate to severe postoperative pain.
3. Be American Society of Anesthesiology (ASA) physical class 1 or 2.
4. Be able to understand the pain intensity evaluation methods.
5. 18kg/m^2<body mass index ≤30 kg/m^2.
6. Female Participants must not be pregnant or lactating. Participants(including their partners)must agree to use appropriate contraception from the time of signing the informed consent form until 3 months after the last dose.No plans for sperm or egg donation during the study period.
7. Be able to understand the study purpose and procedures, agree to participate in the study program, Voluntarily provide written informed consent.

Exclusion Criteria:

1. Have a known allergy to meloxicam or any excipient of meloxicam, aspirin, other non-steroidal anti-inflammatory drugs (NSAIDs) or to any peri- or postoperative medications used in this study.
2. Have a history or clinical manifestations of significant cerebrovascular, respiratory, renal, hepatic, endocrine, neurological, psychiatric systemic diseases, or advanced malignant tumors, and judged by the investigator as unsuitable for participation in this study.
3. Have a history of migraine, anxiety,seizures, cognitive dysfunction, or other psychiatric or neurological disorders that the investigator believes may interfere with the study evaluation.
4. Participants with the following cardiovascular diseases or history:

   1. Severe cardiovascular diseases, NYHA heart function class II or above, myocardial infarction, angina, or coronary artery bypass grafting (CABG) within the preceding 12 months, severe arrhythmias, or abnormal ECG during the screening period judged by the investigator as unsuitable for participation in this study.
   2. Resting systolic blood pressure ≥160mmHg in a sitting or lying position, and/or diastolic blood pressure ≥100mmHg during the screening period, from the signing of the informed consent to before anesthesia induction.
   3. Clinically significant respiratory insufficiency, hypotension, bradycardia occurring intraoperatively or postoperatively before randomization, judged by the investigator as unsuitable for participation in this study.
5. Have another painful physical condition judged by the investigator that may confound the assessments of post operative pain.
6. Have (within 12 months) gastrointestinal ulceration, erforation, gastrointestinal bleeding, or abdominal surgery before the screening period judged by the investigator as unsuitable for participation in this study.
7. Have a known bleeding disorder or be taking agents affecting coagulation judged by the investigator as unsuitable for participation in this study.
8. Participants at high risk of bleeding, including those with congenital bleeding disorders (e.g., hemophilia), thrombocytopenia (platelet count below 0.75× the lower limit of normal), or abnormal platelet function (e.g., idiopathic thrombocytopenic purpura, disseminated intravascular coagulation, congenital platelet dysfunction).
9. ALT or AST >2 ULN, TBIL >1.5 ULN, PT >ULN+3s, APTT ≥ULN+10s, Cr ≥1.5×ULN during the screening period, or any laboratory abnormalities judged by the investigator at screening and/or before surgery that may increase the risk of participation.
10. Blood glucose ≥11.1mmol/L from the screening period to before anesthesia induction.
11. Use of the following drugs (not exceeding 5 half-lives of the drug) before randomization, except for anesthetics and sedative/analgesic drugs used preoperatively for invasive examinations as allowed by the protocol: NSAIDs (including compound preparations containing NSAIDs), opioids, anesthetics, sedatives, hypnotics, anticonvulsants, antipsychotics, other central nervous system inhibitors with analgesic effects, and glucocorticoids (excluding topical and inhaled medications).
12. Use traditional Chinese medicines or proprietary Chinese medicines that could interfere with the evaluation of efficacy or safety judged by the investigator.
13. Have been receiving or have received opioid therapy defined Long-term use (continuous use ≥3 days) of opioid analgesics within 14 days before the screening period.
14. Have a history of alcohol abuse (regularly drinks > 14 units of alcohol per day: 1 unit = 360mL beer or 45mL of 40 % spirits or 150mL wine) within the past 2 years or a history of acute alcohol intoxication, alcohol dependence, drug abuse.
15. Have received any drug/device clinical trials within 3 months before dosing with study medication.
16. Have other conditions that make the subject unsuitable for participation in the clinical study in the opinion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Summed Pain Intensity Difference Over the First 24 Hours (SPID24) | 24 Hours
  Pain intensity was recorded using a Numeric Pain Rating Scale (Range 0-10) where 0 equates to no pain (better), and 10 equates to the worst pain imaginable (worse). Pain intensity scores were to be recorded at the following time points: 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 14 hours, 16 hours, 18 hours and 24 hours post Dose1. Pain intensity differences from baseline at each time point were calculated and a time weighted summed pain intensity difference (SPID) was then calculated. Time weighted SPID calculations were computed by multiplying a weight factor to each score prior to summation. The weight factor at each time point was the time elapsed since the previous observation. A smaller SPID value (i.e. more negative) was better.

SECONDARY OUTCOMES:
Proportion of Participants Utilizing Rescue Analgesia | 48 Hours
  Rescue analgesia (Morphine Hydrochloride Injection 2mg) was available to Participants with inadequately controlled pain upon request.
Number of Doses of Rescue Analgesia Utilized Subject | 48 Hours
  Rescue analgesia (Morphine Hydrochloride Injection 2mg) was available to Participants with inadequately controlled pain upon request.
Number of Times of Rescue Analgesia Utilized Subject | 48 Hours
  Rescue analgesia (Morphine Hydrochloride Injection 2mg) was available to Participants with inadequately controlled pain upon request.
Summed Pain Intensity Difference (SPID) at Other Intervals | 48 Hours
  Pain intensity was recorded using a Numeric Pain Rating Scale (Range 0-10) where 0 equates to no pain (better), and 10 equates to the worst pain imaginable (worse). Pain intensity scores were to be recorded at the following time points: 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 14 hours, 16 hours, 18 hours hours post Dose1. Thereafter pain assessments were to be recorded every 6 hours until 48 hours post Dose 1. Pain intensity differences from baseline at each time point were calculated and a time weighted summed pain intensity difference (SPID) was then calculated. Time weighted SPID calculations were computed by multiplying a weight factor to each score prior to summation. The weight factor at each time point was the time elapsed since the previous observation. A smaller SPID value (i.e. more negative) was better.
TOTPAR (Total Pain Relief) | 48 Hours
  Pain relief will be evaluated considering the Sum of Total Pain Relief (TOTPAR) over 0-12 hours，0-18 hours，0-24 hours，0-48 hours post-dose. Pain relief will be evaluate using a Categorical Pain Relief Rating Scale (0 = No relief, 1 = Mild relief, 2 = Moderate relief, 3 = Marked relief, 4 = complete relief)
Time to First Dose of Rescue Analgesia | 48 Hours
  Rescue analgesia (Morphine Hydrochloride Injection 2mg) was available to Participants with inadequately controlled pain upon request.
Investigator and subject satisfaction scores for analgesic treatment | 48 Hours
  Satisfaction scores will be evaluate using a 5 point scale (0-4) with categories of 0-poor, 1-fair, 2-good, 3-very good, or 4-excellent.

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Cangzhou People's Hospital, Cangzhou
  - The Third Xiangya Hospital Of Central South University, Changsha
  - Heping Hospital Affiliated To Changzhi Medical College, Changzhi
  - Sichuan Academy of Medical Sciengces & Sichuan Provincial People's Hospital, Chengdu
  - The Second People's Hospital Of Chengdu, Chengdu
  - The Third People's Hospital Of Chengdu, Chengdu
  - The First People's Hospital Of Guangyuan, Guangyuan
  - The First affiliated Hospital Of Jinan University, Guangzhou
  - The Affiliated Hospital Of Guizhou Medical University, Guizhou
  - Haikou People's Hospital, Haikou
  - The Second Hospital Of Anhui Medical University, Hefei
  - The First Affiliated Hospital Of University Of South ChinaThe First Affiliated Hospital Of University Of South China, Hengyang
  - Meihekou Central Hospital, Meihekou
  - Nanjing Women and Children's Healthcare Hospital, Nanjing
  - The Second Nanning People's Hospital, Nanning
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The First Affiliated Hospital Of Xi'an Medical University, Xi'an